CLINICAL TRIAL: NCT03509831
Title: A Randomized, Open-label, Crossover Clinical Study to Assess the Safety and the Pharmacokinetic Characteristics of INT-2150 After Oral Administration to Healthy Adult Male Subjects
Brief Title: [KJ-INT-002] BE Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kukje Pharma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KJ-INT-002
Record Dates: First submitted 2018-04-05; First posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Gastritis
MeSH Terms: conditions — Gastritis | interventions — irsogladine; Nizatidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INT2150-A (Other)
  Interventions: Drug: INT-2150; Drug: Irsogladine maleate 2 mg+Nizatidine 150 mg
- INT2150-B (Other)
  Interventions: Drug: INT-2150; Drug: Irsogladine maleate 2 mg+Nizatidine 150 mg

INTERVENTIONS:
Drug: INT-2150 — 1. Period: INT-2150
  2. Period: Irsogladine maleate 2 mg+Nizatidine 150 mg
Drug: Irsogladine maleate 2 mg+Nizatidine 150 mg — 1. Period: Irsogladine maleate 2 mg+Nizatidine 150 mg
  2. Period: INT-2150

SUMMARY:
Assess the Safety and the Pharmacokinetic Characteristics of INT-2150 after Oral Administration to Healthy Adult Male Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Male aged between 19 and 45 years of age inclusive, at the time of signing the informed consent.
2. Body weight >= 50 kilogram (kg) and body mass index within the range 18 - 29.0kg/m^2 (inclusive).
3. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
4. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

1. Patients with a history of abnormal digestive organ, kidney, respiratory, neuroendocrine, cardiovascular, hemato-oncology, urinary, muscloskeletal, immune, the nose and ears, psychiatry, stomach system.
2. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator contraindicates their participation.
3. Systolic blood pressure ≥ 150 or ≤ 100 mmHg, Diasolic blood pressure ≥ 95 or ≤ 55 mmHg.
4. Gastrointestinal disease or with gastrointestinal surgical history which can affect the absorption of the investigational product.
5. Alanine aminotransferase, alkaline phosphatase <=2x upper limit of normal (ULN) total bilirubin > 2.0mg/dl and eGRF <60mL/min/1.73m2
6. History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >21 units for males. One unit is equivalent to 10 gram of alcohol.
7. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days of the biological effect of the investigational product (whichever is longer).

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
AUCt | One day
  Pharmacokinetic Characteristics
Cmax | One day
  Pharmacokinetic Characteristics

SECONDARY OUTCOMES:
AUC∞ | One day
  Pharmacokinetic Characteristics
tmax | One day
  Pharmacokinetic Characteristics
t1/2 | One day
  Pharmacokinetic Characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Heon Cho, Principal Investigator — Inha University Hospital
Locations (1):
- Kukje Pharm, Seongnam-si, South Korea

IPD SHARING:
Plan to Share IPD: Undecided